CLINICAL TRIAL: NCT05901480
Title: An Investigator Initiated Study Evaluating the Safety, Tolerability, and Efficacy of OTOV101N+OTOV101C Injection in Treating Patients With OTOF Mutation-related Deafness
Brief Title: An Investigator Initiated Study for OTOV101N+OTOV101C Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Otovia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTOV101-IIT-101
Record Dates: First submitted 2023-05-09; First posted 2023-06-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-08

CONDITIONS: DFNB9

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients with OTOF mutation-related deafness
  Interventions: Genetic: OTOV101N+OTOV101C Injections

INTERVENTIONS:
Genetic: OTOV101N+OTOV101C Injections — The gene therapy of OTOV101N+OTOV101C injection via intracochlear injection.

SUMMARY:
This study is an investigator initiated study to evaluate the safety, tolerability, and efficacy of OTOV101N+OTOV101C injection in treating patients with OTOF mutation-related deafness. The enrolled subjects who meet the inclusion and exclusion criteria will receive the gene therapy of OTOV101N+OTOV101C injection via intracochlear injection. All participants will return to the hospital for safety and efficacy evaluations at predetermined time points defined by protocol during the study (Week 1 ± 1 Day, Week 2 ± 3 Days, Week 3 ± 3 Days, Month 1 ± 3 Days, Month 2 ± 3 Days, Month 4 ± 6 Days, Month 6 ± 6 Days, Month 9 ± 6 Days, Month 12 ± 6 Days/EOS (end of study)/unscheduled visit).

DETAILED DESCRIPTION:
This study is an investigator initiated study to evaluate the safety, tolerability, and efficacy of OTOV101N+OTOV101C injection in treating patients with OTOF mutation-related deafness.

Subjects who are successfully enrolled will visit the hospital on Day -3 to initiate the glucocorticoid treatment, then be hospitalized on Day -3~-1 to prepare for inner ear gene therapy. On the day of surgery (Day 0), subjects will undergo intracochlear injection of gene therapy products after skin preparation and disinfection of the surgical area and general anesthesia. The round window will be exposed through the tympanic membrane route. Each subject will receive adeno-associated virus (AAV) injection at a dose of 15~30μL of each AAV, mixed at 1: 1 ratio with total volume of 30~60 μL/ear. For subjects without any cochlear implantation, bilateral or unilateral intracochlear injection could be conducted as decided by investigators. For intracochlear injection, the investigators will decide if the second intracochlear injection should be conducted based on dose of the first injection by considering anatomical structure of artificial cochlea and drug loss. The timing of the second injection will be decided by recovery status of the first injection. Subjects will be in hospital for 3 days for observation after receiving the intracochlear injection or follow the routine hospitalization timing of diagnosis/treatment of site, then be discharged after recovery from the surgical operation and receive 1 year follow-up visits.

All subjects will return to the hospital (except in case of non-resistance) for safety and efficacy assessments during the study at the established time points in the protocol (Week 1 ± 1 Day, Week 2 ± 3 Days, Week 3 ± 3 Days, Month 1 ± 3 Days, Month 2 ± 3 Days, Month 4 ± 6 Days, Month 6 ±6 Days, Month 9 ± 6 Days, Month 12 ± 6 Days/EOS (end of study)/Unscheduled) unless encountering force majeure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 years old at the time of signing the informed consent form (ICF); both male and female are eligible.
2. Diagnostic criteria for OTOF-related hearing loss are:

   1. The hearing test and auditory brainstem response (ABR) examination show the presence of hearing loss (based on the testing report conducted within one month prior to signing the informed consent form).
   2. Genetic testing confirms the presence of OTOF gene homozygous or compound heterozygous mutations.
3. Hearing loss: severe (65 dB ≤ hearing threshold < 80 dB) or profound (80 dB ≤ hearing threshold < 95 dB) or total (hearing threshold ≥ 95 dB) hearing loss in both ears (If the testing result of ABR is "waveform is not obtained", the subjects with bilateral hearing threshold <65 dB will be enrolled as determined by the investigator).
4. Vital signs, physical examination, laboratory tests (including whole blood count, blood biochemistry, urinalysis, coagulation function, etc.), and 12-lead electrocardiogram are all normal, or any abnormalities judged by the investigator are clinically non-significant.
5. The subjects and their guardians sign the informed consent form.

Exclusion Criteria:

1. Subjects who have had a severe allergic reaction (NCICTCAE5.0 ≥ 3 Grade) to any drug or its components used in this study in the past;
2. Subjects who have received any gene therapy in the past, or have high levels of neutralizing antibodies (>1:128) in their blood;
3. Subjects who have systemic diseases or are receiving related treatments that may affect hearing or surgical operations;
4. Subjects who cannot tolerate anesthesia;
5. Subjects with inner ear malformations;
6. Subjects who have undergone bilateral cochlear implantation or have a history of major inner ear surgery (as determined by the investigator)(not include unilateral cochlear implantation);
7. Subjects with other genetic mutations causing deafness that may affect the effectiveness of OTOF gene therapy;
8. Subjects with Meniere's disease;
9. Subjects who routinely use ototoxic drugs for other medical conditions;
10. Subjects with congenital deafness caused by non-genetic factors related to birth;
11. Subjects who are currently receiving or may receive immunosuppressive therapy other than this study;
12. Subjects who are allergic or intolerant to glucocorticoid treatment;
13. Subjects with a history of malignant tumors or meningitis;
14. Subjects with a persistent or active infection, positive for hepatitis B surface antigen (HBsAg) with peripheral blood HBV DNA titers higher than the detection limit, positive for hepatitis C virus (HCV) antibodies with peripheral blood HCV RNA titers higher than the detection limit, positive for human immunodeficiency virus (HIV) antibodies, or with other immune deficiency diseases, or positive for syphilis;
15. Subjects of childbearing potential who refuse to take effective contraceptive measures (hormonal or barrier methods or abstinence) from the time of signing the informed consent form until 12 months after receiving AAV injection;
16. Female subjects of childbearing age who have a positive blood pregnancy test result, or are currently pregnant or breastfeeding;
17. Subjects who have participated in any other clinical trial and have received treatment or medication within 4 weeks prior to the first administration (excluding non-interventional studies);
18. Subjects who are unwilling or unable to comply with this study protocol;
19. Subjects whom the investigator believes are unable to participate in this study due to any medical condition or who are unable to complete the follow-up study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-12-06 (Estimated); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to 12 months after unilateral cochlear injection
  Incidence and severity of AEs are assessed by NCI-CTCAE 5.0.
Drug-relatedness of adverse events (AEs) | Up to 12 months after unilateral cochlear injection
  Drug-relatedness of AEs include definitely relevant, probably relevant, possible relevant, possible irrelevant, and definitely irrelevant.
Safety assessment by physical examination | Up to 12 months after unilateral cochlear injection
  Number and percentage of participants with abnormal physical examination findings with clinical significance.
Safety assessment by whole blood count | Up to 12 months after unilateral cochlear injection
  Number and percentage of participants with abnormal laboratory test results (whole blood count) with clinical significance.
Safety assessment by urinalysis | Up to 12 months after unilateral cochlear injection
  Number and percentage of participants with abnormal laboratory test results (urinalysis) with clinical significance.
Safety assessment by blood biochemistry testing | Up to 12 months after unilateral cochlear injection
  Number and percentage of participants with abnormal laboratory test results (blood biochemistry testing) with clinical significance.
Safety assessment by coagulation function testing | Up to 12 months after unilateral cochlear injection
  Number and percentage of participants with abnormal laboratory test results (coagulation function) with clinical significance.
Safety assessment by vital signs | Up to 12 months after unilateral cochlear injection
  Number and percentage of participants with abnormal vital signs with clinical significance.
Safety assessment by electrocardiogram | Up to 12 months after unilateral cochlear injection
  Number and percentage of participants with abnormal ECG readings with clinical significance.
Safety assessment by cranial MRI (Magnetic Resonance Imaging) | Up to 12 months after unilateral cochlear injection
  Changes in cranial MRI relative to baseline, to observe possible signs of infection after gene therapy on inner ear. The MRI conduction is decided by investigator.
Safety assessment by neutralizing antibodies in peripheral blood | Up to 12 months after unilateral cochlear injection
  Changes in neutralizing antibodies relative to baseline in peripheral blood collections. Concentrations of neutralizing antibodies are analyzed by cell-mediated assay in vitro.
Safety assessment by Adeno-Associated Virus (AAV) in peripheral blood | Up to 12 months after unilateral cochlear injection
  Changes in AAV signals relative to baseline in peripheral blood collections. AAV signals are analyzed by real-time PCR assay in vitro.
Safety assessment by CT (Computed Tomography) | Up to 12 months after unilateral cochlear injection
  Changes in cranial CT relative to baseline, to observe possible signs of infection after gene therapy on inner ear. The CT conduction is decided by investigator.

SECONDARY OUTCOMES:
Efficacy assessment by Behavioral audiometry testing | Up to 12 months after unilateral cochlear injection
  Changes in hearing assessment by behavioral audiometry relative to baseline, to observe the improvement of hearing functions after gene therapy on inner ear. Behavioral audiometry assessments are to measure the hearing threshold at different frequencies (pitches) after treatment compared to its baseline values.
Efficacy assessment by ABR (Auditory Brainstem Response) testing | Up to 12 months after unilateral cochlear injection
  Changes in hearing assessment by ABR relative to baseline, to observe the improvement of hearing functions after gene therapy on inner ear. ABR assessments are to measure the electrical response evoked by acoustic stimuli as sound signal is processed along the auditory pathway. Mean ABR air and bone conduction threshold are assessed.
Efficacy assessment by ASSR (Auditory Steady-state Response) testing | Up to 12 months after unilateral cochlear injection
  Changes in hearing assessment by ASSR relative to baseline, to observe the improvement of hearing functions after gene therapy on inner ear. ASSR assessments are to measure the Steady-State electroencephalic response evoked by acoustic stimuli as sound signal is processed along the auditory pathway. Mean ASSR air and bone conduction threshold are assessed.
Efficacy assessment by DPOAE (Distortion Product Otoacoustic Emission) testing | Up to 12 months after unilateral cochlear injection
  Changes in hearing assessment by DPOAE relative to baseline, to observe the improvement of hearing functions after gene therapy on inner ear. DPOAE is defined as sound generated within the cochlear by stimulating the ear with two simultaneous tones of different frequency. DPOAEs serve as an objective measure of hearing sensitivity. Tones will be played from low to high frequencies at soft to moderate levels to assess responses at different regions of the inner ear. DP levels will be recorded for each frequency and ear. Higher DP levels indicate more sensitive hearing. Change from baseline values will be calculated as the reported DP level value minus the baseline value. A negative change from baseline indicates less sensitive hearing.
Efficacy assessment by CM (Cochlear Microphonic) potential | Up to 12 months after unilateral cochlear injection
  Changes in hearing assessment of CM potentials relative to baseline, to observe the improvement of hearing functions after gene therapy on inner ear. CM potentials are measured by Cochlear Response Telemetry System.
Efficacy assessment by tympanometry | Up to 12 months after unilateral cochlear injection
  Changes in hearing assessment of tympanometry relative to baseline, to observe the improvement of hearing functions after gene therapy on inner ear. Tympanometry are used to assess the mobility of the eardrum. Compliance, middle ear pressure and ear canal volume will be recorded and checked to measure function of middle ear and eustachian tube.

CONTACTS AND LOCATIONS:
Overall Officials: Shanzhong Zhang, MD PhD, Study Director — Otovia Therapeutics
Locations (23):
- China (23):
  - Shandong Second Provincial General Hospital, Jinan, Shandong
  - Beijing Tongren Hospital, Beijing
  - Beijing Union Hospital, Beijing
  - Chinese PLA Genreal Hospital, Beijing
  - The Third Bethune Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People Hospital, Chengdu
  - Chongqing Municipal People Hospital, Chongqing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangdong Provincial People Hospital, Guangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of USTC, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Yunnan Provincial First People Hospital, Kunming
  - Dongnan University Zhongda Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - The Second Hospital of Ningbo, Ningbo
  - Shengjing Hospital Of China Medical University, Shenyang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Xijing Hospital, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi J, Zhang L, Lu L, Tan F, Cheng C, Lu Y, Dong W, Zhou Y, Fu X, Jiang L, Tan C, Zhang S, Sun S, Song H, Duan M, Zha D, Sun Y, Gao X, Xu L, Zeng FG, Chai R. AAV gene therapy for autosomal recessive deafness 9: a single-arm trial. Nat Med. 2025 Sep;31(9):2917-2926. doi: 10.1038/s41591-025-03773-w. Epub 2025 Jul 2. PMID 40603731